CLINICAL TRIAL: NCT00004485
Title: Phase I/II Study of Induction of Stable Mixed Chimerism After Bone Marrow Transplantation From HLA-Identical Donors in Children With Sickle Cell Disease
Brief Title: Bone Marrow Transplantation in Treating Children With Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/14243; FHCRC-1373.00
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-09

CONDITIONS: Sickle Cell Anemia
Keywords: genetic diseases and dysmorphic syndromes; hematologic disorders; rare disease; sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases | interventions — Cyclosporine; fludarabine; Mycophenolic Acid; Bone Marrow Transplantation

INTERVENTIONS:
Drug: cyclosporine
Drug: fludarabine
Drug: mycophenolate mofetil
Procedure: Bone Marrow Transplantation

SUMMARY:
RATIONALE: Sickle cell disease is an inherited disorder in which abnormal, crescent-shaped red blood cells interfere with the ability of the blood to carry oxygen through the body and can cause severe pain, stroke, and organ damage. Bone marrow transplantation, is a procedure in which the soft, sponge-like tissue in the center of bones producing white blood cells, red blood cells, and platelets is replaced by bone marrow from a another person. Bone marrow transplantation may be an effective treatment in relieving the symptoms of sickle cell disease.

PURPOSE: Phase I/II trial to study the effectiveness of bone marrow transplantation in treating children who have sickle cell disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a multicenter study. Patients undergo total body irradiation on day 0, followed by allogeneic bone marrow transfusion. Patients also receive fludarabine IV daily and cyclosporine IV twice a day on days -1 to 1. Patients then receive oral cyclosporine on days 1-90, and oral mycophenolate mofetil twice a day on days 0-27.

Patients are followed for 100 days, monthly for 6 months and then annually for 2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of sickle cell anemia with clinically severe disease manifestations defined by: Recurrent painful events (at least 2 painful events in past year) which cannot be explained by other causes Pain lasts at least 4 hours Requires treatment with parenteral narcotics, equianalgesic dose of oral narcotics, or parenteral nonsteroidal antiinflammatory drugs Acute chest syndrome (ACS) with at least 2 episodes within past 2 years that required hospitalization, oxygen, and RBC transfusion Any combination of painful events and ACS episodes that total 2 events within the past year Abnormal cerebral MRI, abnormal angiography (MR or conventional), and abnormal neuropsychologic testing performance

No stage III or IV sickle cell lung disease

Genotypically HLA identical sibling donor available

--Prior/Concurrent Therapy--

No prior transfusions with greater than 5 units RBC

--Patient Characteristics--

Performance status: Karnofsky 70-100%

Hepatic:

* No active hepatitis
* No moderate/severe portal fibrosis

Renal: Glomerular filtration rate at least 30% predicted for age

Neurologic:

* No severe residual functional neurologic impairment
* Hemiplegia alone allowed

Other:

* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 1999-12; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Walters, Study Chair — Children's Hospital of Oakland
Locations (2):
- United States (2):
  - Children's Hospital of Oakland, Oakland, California
  - Fred Hutchinson Cancer Research Center, Seattle, Washington